CLINICAL TRIAL: NCT03757403
Title: RDD1609 as a Treatment for Idiopathic Pruritus Ani: A Randomized Double Blinded Placebo Controlled Crossover Study
Brief Title: RDD1609 as a Treatment for Idiopathic Pruritus Ani
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RDD123
Record Dates: First submitted 2018-11-25; First posted 2018-11-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Idiopathic Pruritus Ani
MeSH Terms: interventions — Mebendazole

STUDY DESIGN:
Intervention Model Description: phase 2a randomized double-blinded placebo-controlled cross-over
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDD1609 followed by Placebo (Experimental): Application on the perianal area BID
  Interventions: Drug: RDD1609; Drug: Mebendazole 100 MG
- Placebo followed by RDD1609 (Experimental): Application on the perianal area BID
  Interventions: Drug: RDD1609; Drug: Mebendazole 100 MG

INTERVENTIONS:
Drug: RDD1609 — RDD1609 to be applied on the perianal area BID
Drug: Mebendazole 100 MG — Mebendazole 100 mg single dose (single prophylactic dose of the anthelmintic medicine)
  Other Names: Vermox

SUMMARY:
This is a double-blind, randomized, placebo-controlled, crossover trial, to test the hypothesis that RDD1609 is effective in treating idiopathic pruritus ani.

DETAILED DESCRIPTION:
This is a phase 2a randomized double-blinded placebo-controlled cross-over design study in patients with idiopathic pruritus ani. 24 patients, male and females, aged 18 -65 with severe idiopathic pruritus ani (VAS score above 60), will be randomized to this study.

Patients that meet all inclusion criteria and do not have exclusion criteria at randomization visit will be randomly assigned to one of the two treatment groups:

Group 1 will receive 3 weeks of RDD1609 for 3 weeks, followed by 3 weeks of treatment with placebo.

Group 2 will receive 3 weeks of treatment with placebo followed by 3 weeks of treatment with RDD1609.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Male and female patients, age 18 - 65 years with idiopathic PA.
3. Screening VAS for itching of 60 mm and above.
4. Female subjects of child-bearing potential must have a negative urine pregnancy test. Females of childbearing potential must practice a highly effective method of pregnancy prevention (defined as <1% pregnancies per 100 women per year) from one month before screening to one month after the follow-up visit, such as: surgical sterilization, hormonal implant, intrauterine device, or male condom + female diaphragm + vaginal spermicide. Female subject with any of the following circumstances is not required to use a highly effective method of pregnancy prevention: status post-hysterectomy; or, status post-tubal ligation; or, post-menopausal state (defined as >= 12 months of spontaneous amenorrhea) or < 12 months of spontaneous amenorrhea with a blood follicle stimulating hormone > 40 MIU/ml.
5. Subject has normal (or abnormal and clinically insignificant) laboratory values at Screening.
6. Subject has the ability to understand the requirements of the study and a willingness to comply with all study procedures.
7. Subject has not used and agrees to abstain from taking any prescription or non-prescription medications, cosmetics, including herbal and dietary supplements (such as St. John's wort) within 7 days prior to the first dose of study medication (unless authorized by the Investigator and Medical Monitor).

Exclusion Criteria:

1. Known hypersensitivity to RDD1609.
2. Known hypersensitivity to Mebendazole.
3. Previously treated with methylene blue for pruritus ani.
4. Randomization VAS for itching that is <25 mm than the screening VAS.
5. Anorectal conditions such as malignant tumors of the anus and rectum, inflammatory bowel disease, fistulain- ano, fissure-in-ano, incontinence, condylomata, and second- and third-degree hemorrhoids and any other anorectal conditions that requires medicinal treatment.
6. Patients who had previous major proctological surgery.
7. Generalized skin disorders.
8. Active psychiatric disorders.
9. Diabetes mellitus all types.
10. Known to be HIV positive.
11. Current or within the last 4 weeks steroid or pregabalin or gabapentin or antihistamine systemic or local treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for itching | 3 weeks
  Change in severity of itch, measured using Visual Analogue Scale score for itching from baseline through the end of treatment. The Visual Analogue Scale is a 10-cm long line (oriented horizontally), on which patients indicate the severity of their itching by crossing the line at the point that corresponded to their itching severity. The left end of the line indicates "no itch" and right end of the line indicates "worth itch ever".
Pruritus Ani Severity Index score | 3 weeks
  Effect of RDD1609 on the Pruritus Ani Severity Index score (Mild, Moderate, Severe, Chronic), which is a grading system used to describe severity of physical findings in patients with pruritus ani.

SECONDARY OUTCOMES:
Safety and Tolerability of RDD1609 ( the frequency of adverse events and serious adverse events) | 3 weeks
  Will be based primarily on the frequency of adverse events and serious adverse events. Other safety data will be summarized as appropriate.

OTHER OUTCOMES:
Dermatology Life Quality Index | 3 weeks
  Effect of treatment on Dermatology Life Quality Index.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Barak, MD, Study Chair — RDD Pharma Ltd; Jeanette Melrose, MD, Principal Investigator — THE ATHERSTONE SURGERY
Locations (4):
- United Kingdom (4):
  - The Atherstone Surgery, Atherstone
  - University Hospitals Bristol NHS Foundation Trust- Location Bristol Royal Infirmary, Bristol
  - Kings Medical Centre, Buckhurst Hill
  - Sheepcot Medical Centre, Watford